CLINICAL TRIAL: NCT02335099
Title: Randomized, Placebo-controlled, Single Blind, Trial to Determine the Safety and Efficacy of Ticagrelor for Maintaining Patency of Arterio-Venous Fistulae Created for Hemodialysis
Brief Title: Determine the Safety/Efficacy of Ticagrelor for Maintaining Patency of Arterio-Venous Fistulae Created for Hemodialysis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Emaad Abdel-Rahman, MD, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17224
Record Dates: First submitted 2014-12-19; First posted 2015-01-09 (Estimated); Results first posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-05

CONDITIONS: End Stage Renal Disease; Vascular Access Patency
Keywords: hemodialysis; vascular access; vascular access patency; ticagrelor; brilinta
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ticagrelor (Active Comparator): 90 mg of ticagrelor to be given orally twice a day for 6 months
  Interventions: Drug: ticagrelor
- Placebo (Placebo Comparator): Placebo drug to be given twice a day for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ticagrelor — ticagrelor 90 mg twice a day for 6 months
  Other Names: Brilinta
  Arms: ticagrelor
Drug: Placebo — 1 pill twice a day for 6 months
  Arms: Placebo

SUMMARY:
This study is a randomized, placebo-controlled, single blind clinical trial. Seventy patients with ESRD on chronic HD and a functioning AVF will be recruited. The following data will be documented on each patient: 1-Age/gender/race/body weight/cause of ESRD 2-Vintage of HD 3-Time since access was placed 4-Type and place of access and blood flow rate of access 5-History of prior access problems 6-Comorbid conditions (Hypertension, coronary artery disease, Diabetes Mellitus, Bleeding problems, peripheral vascular disease). 7-Current medications (Coumadin, Erythropoiesis stimulating agents, heparin, other antiplatelets, digoxin, statins). Patients will be randomized into two groups to receive: Group 1: Ticagrelor 90 mg PO BID Group 2: Placebo drug PO BID.

DETAILED DESCRIPTION:
This study is a randomized, placebo-controlled, single blind clinical trial. Seventy patients with ESRD on chronic HD and a functioning AVF will be recruited. Consent form will be obtained. History and physical, dialysis parameters and laboratory data (CBC, CMP, PTT & INR) will be obtained throughout the study. The following data will be documented on each patient: 1-Age/gender/race/body weight/cause of ESRD 2-Vintage of HD 3-Time since access was placed 4-Type and place of access and blood flow rate of access 5-History of prior access problems 6-Comorbid conditions (Hypertension, coronary artery disease, Diabetes Mellitus, Bleeding problems, peripheral vascular disease). 7-Current medications (Coumadin, Erythropoiesis stimulating agents, heparin, other antiplatelets, digoxin, statins). Patients will be randomized into two groups to receive: Group 1: Ticagrelor 90 mg PO BID Group 2: Placebo drug PO BID.

Subjects will have a screening visit and if they qualify for the study they will have 18 additional visits. All of these visits will occur while the subjects are at their normal dialysis treatment. Subjects will be randomized to either the Ticagrelor group or the placebo group. Subjects will be on study medication for 6 months then they will have a follow up period off drug for 6 months. Subjects will be seen twice a month while on study medication and once a month in the follow up period. While the subjects are on study medication the study team will assess any side effects of the study medication and put their relation to the study drug at each study visit. The study team will use clinical monitoring as suggested by Beathard (21). The study team will document the subject's adherence to the study, if they are hospitalized and what caused their hospitalization. A monthly intra-access flow will be obtained using ultrasound dilution by transonics as part of standard of care. Any change in the clinical assessment of the access, prolonged bleeding (>20 minutes) after removal of needles, trend of decreasing intra-access blood flow as determined by transonic (> 25% or original flow), or an access flow rate < 400 ml/min, will prompt a referral for a fistulogram. If confirmed stenosis (>50% stenosis of the access diameter) an intervention (angioplasty) will be performed. This intervention is part of the subjects standard of care.

ELIGIBILITY:
Inclusion Criteria:

- Patients on chronic hemodialysis with a functioning arterio-venous fistula

Exclusion Criteria:

* Recent history of bleeding over the last 3 months preceding enrollment
* History of bleeding disorder (hemophilia, Von Willebrandt disease, etc….)
* Recent history of blood transfusion over the last 3 months preceding enrollment
* Recent serious injury or surgery over the last 3 months preceding enrollment
* History of gastro-intestinal ulcers
* Moderate-severe hepatic impairment
* Uncontrolled blood pressure (SBP> 200 or DBP >110) post dialysis
* History of stroke
* Pregnant females-self reported
* Hypersensitivity to Aspirin /antiplatelets
* Subjects using peroral anticoagulants

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia - Hospital West Kidney Center Dialysis, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 10 of 54 consented subjects failed screening and were not assigned to the study arms.
Groups:
- Treatment: 90 mg of Ticagrelor to be given orally twice a day for 6 months
Period: Treatment
Arm/Group | Treatment | Placebo
Started | 22 | 22
Completed | 17 | 17
Not Completed | 5 | 5
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Death | 1 | 0
Not completed — Adverse Event | 1 | 2
Period: Follow-up
Arm/Group | Treatment | Placebo
Started | 17 | 17
Completed | 17 | 16
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Placebo | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (12.4) | 60.8 (10.4) | 58.2 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 14 | 12 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 13 | 24
  White | 6 | 4 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility and Safety of Ticagrelor in Hemodialysis Patients
Description: Number of Participants with prolonged bleeding (>30 minutes) after removal of needles
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 17 | 17
Participants | 1 | 3
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority; p = 0.32, Fisher Exact; Odds Ratio (OR) = 3.77, 95% CI 2-sided [0.27 to 217.52]

2. Secondary Outcome: Treatment Efficacy of Ticagrelor to Preserve Patency of Hemodialysis Vascular Access
Description: Percentage of participants with stenosis free survival
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 17 | 17
percentage of participants | 72.2 [54.2 to 96.2] | 75.0 [56.5 to 99.5]
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority; p = 0.82, Log Rank; Cox Proportional Hazard = 0.86, 95% CI 2-sided [0.23 to 3.20]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 1/17 | 1/17
Serious Adverse Events (participants affected / at risk) | 1/17 | 1/17
Other Adverse Events (participants affected / at risk) | 3/17 | 2/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=17) | Placebo (N=17)
cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=17) | Placebo (N=17)
increased diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
transient ischemic attack - stroke (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
tickling feeling in head (General disorders) | 1 (1) | 0 (0)
bruise on hand (General disorders) | 1 (1) | 0 (0)
bloody drops on penis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
cold (Infections and infestations) | 0 (0) | 1 (1)
worsening pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The results may be affected by the enrollment that did not reach a goal of 70 subjects with only 34 subject or 48.5% of the projected number completing the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/99/NCT02335099/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/99/NCT02335099/ICF_001.pdf